CLINICAL TRIAL: NCT00032292
Title: A Phase I/II, Open-Label, Dose-Escalation, Pilot Study to Evaluate Safety and Preliminary Efficacy of Visilizumab as Primary Therapy for Acute Graft-Versus-Host Disease After Hematopoietic Cell Transplantation
Brief Title: Research Study of Visilizumab for Treatment of Acute Graft Versus Host Disease
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Facet Biotech (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 291-405
Record Dates: First submitted 2002-03-14; First posted 2002-03-18 (Estimated); Last update posted 2012-03-13 (Estimated); Status verified 2012-03

CONDITIONS: Graft vs Host Disease
MeSH Terms: conditions — Graft vs Host Disease | interventions — visilizumab

INTERVENTIONS:
Drug: Visilizumab

SUMMARY:
The purpose of this Phase I/II, open-label, dose-escalation study is to evaluate an investigational monoclonal antibody administered as a first-line therapy to patients with acute, Grade II, III, or IV graft-versus-host disease (GVHD). Patients will be eligible for enrollment within 24 hours of beginning standard steroid treatment. The research is being conducted at up to 10 clinical research sites in the US.

DETAILED DESCRIPTION:
A Phase I/II, open-label, dose-escalation pilot study designed to obtain preliminary safety, pharmacokinetic (PK) and efficacy information on visilizumab administered as a first-line therapy to patients with acute, Grade II, III, or IV graft-versus-host disease (GVHD). It is anticipated that up to 34 patients at up to 10 study centers could be eligible for enrollment in this study. Patients will be eligible for enrollment within 24 hours of beginning standard steroid treatment (2 mg/kg of methylprednisolone IV, or 10 mg/kg hydrocortisone IV, per day). Steroids will be rapidly tapered over one week following visilizumab administration.

ELIGIBILITY:
* Patients who develop Grade II, III, or IV acute GVHD following allogeneic hematopoietic cell transplantation
* Patients receiving GVHD prophylaxis including cyclosporine or tacrolimus
* Clinical findings: skin thickening, joint contraction, oral ulceration, diarrhea.
* Patients with an onset date of acute GVHD that is less than or equal to 100 days posttransplant.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 34
Dates: Start 2002-03; Primary Completion 2006-08 (Actual); Study Completion 2006-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - City of Hope National Medical Center, Duarte, California
  - Stanford University Medical Center, Stanford, California
  - Washington University School of Medicine, St Louis, Missouri
  - Duke University, Durham, North Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - MD Anderson Cancer Center, Houston, Texas
  - Fred Hutchinson Cancer Research Center, Seattle, Washington